CLINICAL TRIAL: NCT02486588
Title: Increasing Engagement With the Vitality HealthyFood Benefit: A Randomized Field Trial Proposal
Brief Title: Increasing Engagement With a Healthy Food Benefit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 822607
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Purchasing Behaviors; Nutrition
Keywords: Financial incentives; Messaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control--no weekly message (No Intervention): 10% cash back level, no weekly message, and the standard monthly message
- General Weekly Message (Experimental): 10% cash back, general weekly message, standard monthly message
  Interventions: Other: Messaging; Other: Financial incentives
- Personalized Weekly Message (Experimental): 10 % cash back, personalized weekly message, standard monthly message
  Interventions: Other: Messaging; Other: Financial incentives
- 25 percent cash back (Experimental): 25% cash back, personal weekly message, standard monthly message
  Interventions: Other: Messaging; Other: Financial incentives
- Standard monthly message (Experimental): 10%+15% cash back, personal weekly message, standard monthly message
  Interventions: Other: Messaging; Other: Financial incentives
- Unbundled monthly message (Experimental): 10%+15% cash back, personal weekly message, unbundled monthly message
  Interventions: Other: Messaging; Other: Financial incentives

INTERVENTIONS:
Other: Messaging — See detailed study description for overview of the different messaging interventions in this study
  Arms: 25 percent cash back; General Weekly Message; Personalized Weekly Message; Standard monthly message; Unbundled monthly message
Other: Financial incentives — See detailed study description for overview of the different financial incentive-based interventions in this study
  Arms: 25 percent cash back; General Weekly Message; Personalized Weekly Message; Standard monthly message; Unbundled monthly message

SUMMARY:
In collaboration with Vitality/Discovery in South Africa, an RCT amongst adult enrolled in the lowest tier of Vitality's HealthyFood benefit will be conducted. We will compare the effect of various messaging, and financial incentive strategies on healthy food purchasing behaviors in this population.

DETAILED DESCRIPTION:
The Vitality HealthyFood benefit is a three-tiered incentive program designed to encourage healthier food choices amongst members of Discovery Health's Vitality program. Once enrolled in the benefit, participating members can receive 10%, 15%, or 25% cash-back on the healthy foods they purchase at selected grocers. And, while overall enrolment in the program is high, there was been difficulty documenting change in purchasing behaviors; healthy foods have remained a consistent 25-30% of food spend, and unhealthy foods at around 15%. In the current study we would like to test whether differing types of messages and financial incentive structures may be more salient and motivating and have a greater impact on food-purchasing decisions. The proposed study will be a collaboration between Discovery Health/Vitality and researchers at the Perelman School of Medicine at the University of Pennsylvania. In the proposed RCT, Vitality members currently enrolled in the lowest tier (10% level) of the HealthyFood will be randomized to various messaging and financial incentive structures. We will then compare the effectiveness of these different interventions at increasing healthy food purchases among enrolled members.

This study will be a randomized field trial of the combination of several theoretically-motivated interventions: varying weekly messaging, financial incentives, and monthly messaging.

Messaging and financial incentives

Weekly Messaging strategies There are three weekly messaging strategies we want to test. The goal of the messages is to increase the salience of the HealthyFood programme for enrolled members. The three strategies were chosen to enable us to compare the impact of no weekly message vs. a general weekly message vs. a tailored weekly message. The messages will be sent via SMS to all subjects and will be delivered on the same day of the week.

No weekly message-A subset of study subjects will receive no weekly SMS message. This is consistent with the current benefit structure.

General weekly message-A subset of study subjects will receive a weekly SMS that provides general information on the HealthyFood programme and on eating a healthier diet.

Personalized (tailored) weekly message-A subset of study subjects will receive a weekly SMS that includes details about their individual purchasing behavior over the past week. This message will highlight both the percentage and item breakdown of their purchases that were healthy vs. unhealthy.

Financial Incentive Structures

There are three different incentive structures we will test in this study. The goal of the financial incentives is to increase members' motivation to purchase healthy foods. Two of the strategies are currently part of the HealthyFood programme, the third is a new structure which introduces a economic disincentive on the purchase of unhealthy foods.

10% cash-back: This is the current cash-back level for all subjects at the start of on the study. This group is included as a comparison for the other incentive structures.

25% cash back: A subset of study subjects will experience an increase in their cash-back percentage from 10% to 25% of healthy food purchases. The purpose of this group is to assess whether the increase from a 10% level to a 25% level of cash-back is sufficiently large to influence purchasing behaviors.

10% + 15% (healthy-unhealthy): A subset of study subjects will become eligible for additional 15% cash-back above their current 10% level. This additional 15% cash-back will be based on the net monetary amount between their healthy and unhealthy purchases. With this structure, an individual will only receive additional cash-back (above the 10%) if they spend more on healthy foods than on unhealthy foods, and will be able to maximize their cash-back rewards by purchasing only healthy foods.

Monthly Messaging Strategies

Currently all Vitality members enrolled in the HealthyFood programme receive a monthly SMS message informing them of their cash-back deposit.

Bundled deposit SMS (standard)-This message will be the same message that Vitality currently sends to members enrolled in the program me.

Unbundled deposit SMS-Given the introduction of a new incentive structure which includes a penalty for unhealthy purchases, we wanted to test a message strategy which increases the salience of these potential financial losses.

By combining these different weekly messages, incentive structures, and monthly message, the study team determined the aforementioned 6 study arms of interest.

ELIGIBILITY:
Inclusion Criteria:

* For this study, we will focus on the following individuals:

  1. Adult members of Vitality Health who have activated their HealthyFood benefit in 2014 but have not completed the Vitality Age calculation or Vitality Healthy Check, and therefore are on a 10% cash- back reward level on healthy food purchases.
  2. Members who have chosen Woolworths as their preferred HealthyFood partner.
  3. Members with an available email address and SMS-capable telephone
  4. Members with meeting specified spending cutoff (R1000 total spend in the previous month, at least 90% of which was spent at Woolworth's.)

Exclusion Criteria:

* Anyone who does not meet all of the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7314 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Buttenheim, Phd, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gopalan A, Shaw PA, Lim R, Paramanund J, Patel D, Zhu J, Volpp KG, Buttenheim AM. Use of financial incentives and text message feedback to increase healthy food purchases in a grocery store cash back program: a randomized controlled trial. BMC Public Health. 2019 May 31;19(1):674. doi: 10.1186/s12889-019-6936-5. PMID 31151390

RESULTS

PARTICIPANT FLOW:
Groups:
- 10% Cash, no Weekly Message, Standard Monthly SMS: 10% cash back level, no weekly message, and the standard monthly message
- 10% Cash, General Weekly SMS, Standard Monthly SMS: 10% cash back, general weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- 10% Cash, Personal Weekly SMS, Standard Monthly SMS: 10 % cash back, personalized weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- 25% Cash, Personal Weekly SMS, Standard Monthly SMS: 25% cash back, personal weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS: 10%+15% cash back, personal weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- 10+15%NET, Personal Weekly SMS, Unbundled Monthly SMS: 10%+15% cash back, personal weekly message, unbundled monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
Period: Overall Study
Arm/Group | 10% Cash, no Weekly Message, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET, Personal Weekly SMS, Unbundled Monthly SMS
Started | 1188 | 1252 | 1220 | 1206 | 1243 | 1205
Completed | 450 | 502 | 465 | 468 | 497 | 459
Not Completed | 738 | 750 | 755 | 738 | 746 | 746
Not completed — Randomized in error- ineligible | 738 | 750 | 755 | 738 | 746 | 746

BASELINE CHARACTERISTICS:
Groups:
- 10% Cash, no Weekly SMS, Standard Monthly SMS: 10% cash back level, no weekly message, and the standard monthly message
- 10% Cash Back, Personal Weekly SMS, Standard Monthly SMS: 10 % cash back, personalized weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- 25% Cash Back, Personal Weekly SMS, Standard Monthly SMS: 25% cash back, personal weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- 10+15%NET Cash, Personal Weekly SMS, Standard Weekly SMS: 10%+15% cash back, personal weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- 10+15%NET Cash, Personal Weekly SMS, Unbundled Monthly SMS: 10%+15% cash back, personal weekly message, unbundled monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
- Total: Total of all reporting groups
Arm/Group | 10% Cash, no Weekly SMS, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash Back, Personal Weekly SMS, Standard Monthly SMS | 25% Cash Back, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Weekly SMS | 10+15%NET Cash, Personal Weekly SMS, Unbundled Monthly SMS | Total
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459 | 2841
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.8) | 48.3 (11.7) | 47 (11.6) | 47.4 (11.6) | 47.7 (11.9) | 48.5 (12) | 47.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 225 | 220 | 207 | 245 | 212 | 1321
  Male | 238 | 277 | 245 | 261 | 252 | 247 | 1520
Household Size [Mean (Standard Deviation); unit: people] | 3 (1.3) | 2.9 (1.3) | 3 (1.2) | 3 (1.2) | 2.9 (1.2) | 2.9 (1.3) | 2.9 (1.2)
Vitality membership length [Mean (Standard Deviation); unit: Weeks] | 110.5 (56.9) | 110.1 (56.2) | 111.7 (58.3) | 107.3 (55.6) | 112.2 (58.2) | 112.4 (57.8) | 110.7 (57.1)
Region [Count of Participants; unit: Participants]
  Gauteng | 289 | 329 | 302 | 326 | 329 | 291 | 1866
  Kwazulu-Natal | 39 | 41 | 46 | 35 | 51 | 43 | 255
  Western Cape | 86 | 102 | 76 | 72 | 83 | 85 | 504
  Other | 36 | 30 | 41 | 35 | 34 | 40 | 216
Shopping trips [Mean (Standard Deviation); unit: trips per month] | 7.9 (4.4) | 7.9 (4.1) | 8.1 (4) | 7.7 (4.3) | 7.9 (4.1) | 8.3 (4.2) | 8 (4.2)
Monthly healthy spending [Mean (Standard Deviation); unit: Rand (South African currency) per month] | 895 (548.9) | 923.4 (608.9) | 851.8 (511.9) | 843.5 (506) | 878.9 (540.5) | 901.1 (521.4) | 883.4 (541.9)
Monthly unhealthy spending [Mean (Standard Deviation); unit: Rand (South African currency) per month] | 558.3 (347.1) | 539 (302.2) | 549 (326.1) | 515 (303.6) | 532 (313) | 526.6 (332.4) | 536.5 (320.6)
Monthly neutral spending [Mean (Standard Deviation); unit: Rand (South African Currency) per month] | 1823.5 (963.5) | 1760.5 (881.9) | 1818.8 (944.6) | 1727.3 (888.4) | 1736.5 (930.6) | 1786.6 (900.5) | 1774.6 (918.1)
Monthly healthy items [Mean (Standard Deviation); unit: Items per month] | 36.1 (21.2) | 37.5 (23.7) | 34.9 (20.5) | 34.8 (21) | 35.9 (21.6) | 37.1 (20.6) | 36.1 (21.5)
Monthly unhealthy items [Mean (Standard Deviation); unit: Items per month] | 26.4 (18.4) | 24.6 (14.9) | 25.2 (15.8) | 23.7 (15.1) | 24.2 (15.4) | 24.1 (16.4) | 24.7 (16)
Monthly neutral items [Mean (Standard Deviation); unit: Items per month] | 53.7 (28.8) | 51.8 (26.2) | 52.8 (27) | 50.2 (25.7) | 50.7 (26.1) | 52.2 (27) | 51.9 (26.8)
Monthly proportion of spending on healthy foods [Mean (Standard Deviation); unit: Percent of spending] | 27.5 (10.4) | 28.3 (11.8) | 26.6 (9.7) | 27.7 (10.2) | 27.9 (10.5) | 28.5 (11.4) | 27.7 (10.7)
Monthly proportion of spending on unhealthy foods [Mean (Standard Deviation); unit: Percent of spending] | 17.8 (7.6) | 17.7 (7.3) | 17.7 (7.6) | 17.3 (6.8) | 17.7 (7.5) | 16.9 (7.5) | 17.5 (7.4)
Monthly proportion of food items that were healthy [Mean (Standard Deviation); unit: Percent of items] | 31.4 (11.2) | 32.5 (12.7) | 30.8 (10.7) | 32.1 (11.3) | 32.2 (11.6) | 33.1 (12.8) | 32 (11.8)
Monthly proportion of food items that were unhealthy [Mean (Standard Deviation); unit: Percent of items] | 22.6 (9.5) | 22.1 (9.3) | 22.5 (9.4) | 21.9 (9) | 22.1 (9.2) | 21.1 (9.3) | 22.1 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Monthly % Healthy Food Expenditure
Description: The difference in monthly healthy food expenditures between arms. This measure is defined as the monthly amount spent on healthy foods divided by the total monthly amount spent on food, multiplied by 100.
  For those individuals who had no recorded expenditure in a given month, they will be assigned 0% healthy food expenditure that month; in this way, this outcome can be considered a composite score of being engaged in the healthy food program (0%=not engaged) and the level of engagement (if monthly expenditure >0). Each individual's data will be averaged across the intervention period.
Time Frame: Monthly over 6 month intervention period
Measure: Mean (Standard Deviation); unit: Percentage of money per month
Groups:
- 10+15% Cash, Personal Weekly SMS, Standard Monthly SMS: 10%+15% cash back, personal weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
Arm/Group | 10% Cash, no Weekly SMS, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
Percentage of money per month | 24.8 (11.4) | 26.8 (12.9) | 24.9 (11.7) | 25.7 (11.5) | 25.9 (12.7) | 26.5 (13)

2. Secondary Outcome: Monthly % Unhealthy Food Expenditure
Description: The difference in monthly unhealthy food expenditures between arms. This measure is defined as the monthly amount spent on unhealthy foods divided by the total monthly amount spent on food, multiplied by 100.
  The average over the full intervention months will be calculated within an individual and compared between arms. To be complementary with the primary endpoint analysis, in a month where an individual is not engaged in the program (0 total monthly expenditure) the worst-score (100) is imputed for that month. A similar MI approach will also be conducted as a sensitivity analysis.
Time Frame: Monthly over 6 month intervention period
Measure: Mean (Standard Error); unit: Percentage of money per month
Groups:
- 10+15%NET, Personal Weekly SMS, Standard Monthly SMS: 10%+15% cash back, personal weekly message, standard monthly message
  Messaging: See detailed study description for overview of the different messaging interventions in this study
  Financial incentives: See detailed study description for overview of the different financial incentive-based interventions in this study
Arm/Group | 10% Cash, no Weekly SMS, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
Percentage of money per month | 24.4 (20.1) | 21.7 (17.2) | 22.4 (17.7) | 21.7 (17.1) | 23.9 (19.9) | 22.3 (19.1)

3. Secondary Outcome: Monthly % Healthy Items
Description: The difference in monthly healthy food items purchased between arms. This measure is defined as the monthly number of healthy food items divided by the total monthly number of food items.
  The average over the full intervention months will be calculated within an individual and compared between arms. To be complementary with the primary endpoint analysis, in a month where an individual is not engaged in the program (0 total monthly expenditure) the worst-score (0) is imputed for that month. A similar MI approach will also be conducted as a sensitivity analysis.
Time Frame: Monthly over 6 month intervention period
Measure: Mean (Standard Deviation); unit: Percentage of items per month
Groups:
- 10% Cash, no Weekly SNS, Standard Monthly SMS: 10% cash back level, no weekly message, and the standard monthly message
Arm/Group | 10% Cash, no Weekly SNS, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
Percentage of items per month | 27.8 (12.5) | 30.2 (13.9) | 28.4 (12.7) | 29.5 (12.8) | 28.9 (13.6) | 30 (14.5)

4. Secondary Outcome: Monthly % Unhealthy Items
Description: The difference in monthly unhealthy food items purchased between arms. This measure is defined as the monthly number of unhealthy food items divided by the total monthly number of food items.
  The average over the full intervention months will be calculated within an individual and compared between arms. To be complementary with the primary endpoint analysis, in a month where an individual is not engaged in the program (0 total monthly expenditure) the worst-score (100) is imputed for that month. A similar MI approach will also be conducted as a sensitivity analysis.
Time Frame: Monthly over 6 month intervention period
Measure: Mean (Standard Deviation); unit: Percentage of items per month
Arm/Group | 10% Cash, no Weekly SMS, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
Percentage of items per month | 29.4 (19.8) | 26.6 (17.5) | 27.2 (17.7) | 26.3 (17.2) | 28.5 (19.8) | 26.9 (19.2)

5. Secondary Outcome: Percentage Change in Monthly % Healthy Food Expenditures Between Arms
Description: Examining the difference in healthy food expenditure trends between arms where the % health food expenditure is defined as describe for outcome 1 (above)
Time Frame: During the 6 month intervention period
Measure: Mean (Standard Error); unit: percentage change in % healthy spending
Arm/Group | 10% Cash, no Weekly SMS, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
percentage change in % healthy spending | -.0839 (.0062) | -.0777 (.0059) | -.0717 (.0061) | -.0769 (.0062) | -.0729 (.0059) | -.0742 (.0062)

6. Secondary Outcome: Percent Change in Monthly %Unhealthy Food Expenditures Between Arms
Description: Examining the difference in unhealthy food expenditure trends between arms where %unhealthy food expenditure is defined as described for Outcome 2 (above).
Time Frame: During the 6 month intervention period
Measure: Mean (Standard Error); unit: Percent change in % unhealthy food spend
Arm/Group | 10% Cash, no Weekly Message, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
Percent change in % unhealthy food spend | .0836 (.0100) | .0679 (.0095) | .0579 (.0099) | .0823 (.0098) | .0928 (.0095) | .0786 (.0099)

7. Secondary Outcome: Percent Change for Monthly % Healthy Food Items Between Arms
Description: Examining the difference in proportion healthy food item trends between arms where % healthy food items is defined as described for Outcome 3 (above)
Time Frame: During the 6 month intervention period
Measure: Mean (Standard Error); unit: Percent change in % healthy food items
Arm/Group | 10% Cash, no Weekly Message, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
Percent change in % healthy food items | -.0753 (.0066) | -.0650 (.0062) | -.0571 (.0064) | -.0659 (.0064) | -.0684 (.0062) | -.0722 (.0065)

8. Secondary Outcome: Percent Change in Monthly %Unhealthy Food Items Between Arms
Description: Examining the difference in proportion unhealthy food item trends between arms where % unhealthy food items is defined as described for Outcome 5 (above).
Time Frame: During the 6 month intervention period
Measure: Mean (Standard Error); unit: Percent change in % unhealthy food items
Arm/Group | 10% Cash, no Weekly Message, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET, Personal Weekly SMS, Unbundled Monthly SMS
Number analyzed (Participants) | 450 | 502 | 465 | 468 | 497 | 459
Percent change in % unhealthy food items | .0896 (.0099) | .0698 (.0094) | .0639 (.0098) | .0854 (.0097) | .1000 (.0094) | .0817 (.0098)

ADVERSE EVENTS:
Arm/Group | 10% Cash, no Weekly SMS, Standard Monthly SMS | 10% Cash, General Weekly SMS, Standard Monthly SMS | 10% Cash, Personal Weekly SMS, Standard Monthly SMS | 25% Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Standard Monthly SMS | 10+15%NET Cash, Personal Weekly SMS, Unbundled Monthly SMS
Serious Adverse Events (participants affected / at risk) | 0/1188 | 0/1252 | 0/1220 | 0/1206 | 0/1243 | 0/1205
Other Adverse Events (participants affected / at risk) | 0/1188 | 0/1252 | 0/1220 | 0/1206 | 0/1243 | 0/1205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No